CLINICAL TRIAL: NCT07268638
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Praliciguat in Patients With Biopsy-Confirmed Focal Segmental Glomerulosclerosis
Brief Title: A Study of Praliciguat in Participants With Focal Segmental Glomerulosclerosis (FSGS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKB-1973-CI-0001
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: Glomerular Disease; Chronic Kidney Disease; Proteinuria; Urine protein-to-creatinine ratio
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Renal Insufficiency, Chronic; Proteinuria | interventions — praliciguat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Praliciguat (Experimental): Praliciguat will be administered daily with dose escalation to a target dose during a 24-week double-blind period, followed by a 24-week open-label treatment period.
  Interventions: Drug: Praliciguat
- Placebo (Placebo Comparator): Matching placebo will be administered daily for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Praliciguat — Oral Tablet
  Arms: Praliciguat
Other: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study designed to evaluate the efficacy and safety of praliciguat in adults with biopsy-confirmed focal segmental glomerulosclerosis (FSGS). Participants will be randomized 1:1 to receive praliciguat or placebo for initial 24 week treatment period. Following this double-blind period, all participants will receive praliciguat in an open-label extension for an additional 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. UPCR ≥1 (g/g) during screening.
2. On maximally tolerated ACEi or ARB per principal investigator discretion within 1 month of informed consent.
3. Estimated glomerular filtration rate ≥25 milliliters per minute per 1.73 square meters by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
4. Kidney biopsy within 3 years of screening consistent with FSGS or documentation of a genetic mutation in a podocyte protein associated with FSGS.

Exclusion Criteria:

1. Collapsing FSGS in the kidney biopsy report.
2. Sickle cell disease.
3. HbA1c >8% or non-fasting blood glucose >180 milligram/decilitre.
4. Uncontrolled hypertension (≥160/100 millimeters of mercury)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in urine protein-to-creatinine ratio (UPCR) | Baseline (Day 1) and up to Week 24

SECONDARY OUTCOMES:
Percentage of Participants with Partial Remission at Week 24 | Up to Week 24
  Partial remission is defined as 40% UPCR reduction and UPCR<1.5 gram/gram (g/g).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Investigator Site #2, Chula Vista, California
  - Investigator Site # 1, Lawrenceville, Georgia
  - Investigator Site #3, Chicago, Illinois
  - Investigator Site #4, Chattanooga, Tennessee
  - Investigator Site #5, Arlington, Texas

IPD SHARING:
Plan to Share IPD: No